CLINICAL TRIAL: NCT01593306
Title: Concurrent Chemoradiotherapy With Weekly Cisplatin Versus Concurrent Chemoradiotherapy With Weekly Cisplatin and Paclitaxel in Locally Advanced Carcinoma Cervix
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indira Gandhi Medical College, Shimla (Other)
Responsible Party: Principal Investigator, Dr Pragyat Thakur, Junior Resident, department of radiotherapy, Principal Investigator, Indira Gandhi Medical College, Shimla
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pragyat1805
Record Dates: First submitted 2012-05-03; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Carcinoma Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — TP protocol; Cisplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cisplatin and paclitaxel with concurrent radiotherapy (Experimental): weekly cisplatin at 30mg/m2 and paclitaxel at 50mg/m2 are given with concurrent radiotherapy at 2Gy per fraction at 5 fractions per week for 5 weeks followed by either low dose rate (LDR) Intracavitary (I/C) Brachytherapy or supplement Chemoradiotherapy (CRT); if not fit for I/C Brachytherapy
  Interventions: Drug: Paclitaxel, Cisplatin
- cisplatin with concurrent radiotherapy (Active Comparator): weekly cisplatin @ 40mg/m2 is given along with concurrent radiotherapy at 2Gy per fraction with 5 fractions per week for 5 weeks followed by LDR I/C brachytherapy or supplement CRT; if not fit for I/C Brachytherapy
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Paclitaxel, Cisplatin — intravenous paclitaxel infusion at 50mg/m2/week and cisplatin at 30mg/m2/week for 5 weeks. if supplement Chemo Radiotherapy is required then similar dose per week for 2 more weeks.
  Arms: cisplatin and paclitaxel with concurrent radiotherapy
Drug: Cisplatin — intravenous infusion of cisplatin 40mg/m2/week for 5 weeks. if I/C Brachytherapy is not feasible then supplement CRT given with similar dose of cisplatin for 2 more cycles.
  Arms: cisplatin with concurrent radiotherapy

SUMMARY:
The purpose of this study is to check whether addition of paclitaxel to cisplatin and radiation therapy will improve the outcome in locally advanced carcinoma cervix.

DETAILED DESCRIPTION:
Carcinoma cervix is the 2nd most common malignancy among females and about 86% of this burden occurs in developing countries. India accounts for 27% of world cervical cancer burden; and most of them are of locally advanced stage ie stage IIA to IVA.

Significant development in radiation techniques and addition of cisplatin based chemotherapy to radiation schedule has led to improved survival but still it is far from satisfactory with 20 to 25% patients failing locally while 10 to 20% patients fail at distant sites. Novel techniques are required to improve this dismal rate.

Thus investigators intended to use combination chemotherapy with paclitaxel and cisplatin, considering that paclitaxel is a taxane which has shown good efficacy in other solid tumors such as ovary, lung and breast; it has also shown radiosensitizing effect in cervical cancer cell lines and it has also been shown to be effective in phase III trials with cisplatin in metastatic and recurrent carcinoma cervix.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven carcinoma cervix
* age 18 years to 65 years
* stage IIA, IIB, IIIA & IIIB according to FIGO 2009

Exclusion Criteria:

* age > 65 years and < 18 years
* stage IA, IB, IVA & IVB
* Histology other than squamous cell, adenocarcinoma or adenosquamous carcinoma
* history of prior pelvic surgery for cancer, prior pelvic radiotherapy or prior chemotherapy.
* deranged renal function test and liver function test
* KPS >= 60
* distant metastasis

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-10 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
clinical response of the disease | up to 1 year
  to compare clinically, the disease response and local control of combination chemotherapy with weekly cisplatin and paclitaxel with concurrent Radiotherapy Vs single agent cisplatin with concurrent Radiotherapy in locally advanced carcinoma cervix

SECONDARY OUTCOMES:
number of patients with adverse events | during treatment, 14 weeks
  to monitor number of treatment related adverse events in both the arms

CONTACTS AND LOCATIONS:
Overall Officials: Pragyat Thakur, MBBS, Principal Investigator — Indira Gandhi Medical College, Shimla
Locations (1):
- Indira Gandhi Medical College, Shimla, Himachal Pradesh, India

REFERENCES:
- [Derived] Thakur P, Seam R, Gupta M, Gupta M. Prospective randomized study comparing concomitant chemoradiotherapy using weekly cisplatin & paclitaxel versus weekly cisplatin in locally advanced carcinoma cervix. Ann Transl Med. 2016 Feb;4(3):48. doi: 10.3978/j.issn.2305-5839.2015.11.19. PMID 26904570